CLINICAL TRIAL: NCT02679885
Title: Assay of Teriflunomide Concentrations in Males Taking Teriflunomide for Treatment of Multiple Sclerosis and Their Female Sexual Partners
Brief Title: Teriflunomide Male Transmission Study
Status: Completed | Type: Observational
Sponsor: Griffin Hospital (Other)
Responsible Party: Principal Investigator, Joseph B. Guarnaccia, Director, Griffin Hospital
Other Study IDs: TERI001
Record Dates: First submitted 2016-02-02; First posted 2016-02-10 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
It is known that teriflunomide, a treatment for relapsing forms of multiple sclerosis, can be found in low concentrations in semen. Because the drug has been associated with teratogenicity in laboratory animals, the question is raised as to whether the drug can be detected in female partners of sexually active males who are taking the drug to treat their multiple sclerosis.

DETAILED DESCRIPTION:
A total of 10 couples were enrolled in the study. Females partners had undetectable or borderline levels of teriflunomide.

ELIGIBILITY:
Inclusion Criteria:

1. Males with relapsing forms of multiple sclerosis appropriately treated with teriflunomide 14 mg po daily;
2. Continuous treatment for three months with good compliance as assessed by the investigator
3. Age between 18 and 55
4. Penile-vaginal intercourse with a female partner at least twice a month with unimpeded ejaculation.
5. Compliance with safety assessments, e.g., regular bloodwork for complete blood count and liver function testing as recommended in the Package Insert
6. Able to give informed consent

Females

1. Regular sexual intercourse with a male partner who is actively taking teriflunomide
2. Age between 18 and 55
3. Able to give informed consent
4. Negative urine pregnancy test at the time of blood sampling
5. Reliable contraception that does not involve barrier methods

Exclusion Criteria:

1. Use of barrier methods of contraception
2. For males, contraindications to the continued use of teriflunomide
3. Couples that are actively trying to conceive
4. For males, noncompliance with teriflunomide therapy
5. Inability or unwilling to give consent or comply with the protocol
6. Pregnancy of the female sexual partner.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants in this study will include approximately twenty heterosexual couples. The male partner will be a subject who has been taking teriflunomide as part of his multiple sclerosis treatment for at least three months and engaging in active sexual relations with his female spouse or partner.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Serum levels of teriflunomide in males and their female partners | Up to one year
  single laboratory evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Guarnaccia, MD, Principal Investigator — MSTC
Locations (1):
- Multiple Sclerosis Treatment Center at Griffin Hospital, Derby, Connecticut, United States